CLINICAL TRIAL: NCT04650412
Title: Integrated Care of Co-morbidities vs Standard Care After Acute Hypercapnic Respiratory Failure in the Intensive Care Unit: a Randomized Controlled Trial
Brief Title: Integrated Care of Co-morbidities vs Standard Care After AHRF in the Intensive Care Unit
Acronym: TMIRA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: delayed recruitment and lack of refinancing
Sponsor: CTU (Other)
Collaborators: Dan Adler is not working anymore at UGeneva, and nobody replaced him. This study is stopped (Unknown)
Responsible Party: Sponsor-Investigator, CTU, Principal investigator, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-01879
Record Dates: First submitted 2020-11-18; First posted 2020-12-02 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Acute Hypercapnic Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial (bundle of comorbidity care vs standard care)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Bundle of comorbidities care
  Interventions: Other: Bundle of comorbidities care
- Control (No Intervention): Standard care

INTERVENTIONS:
Other: Bundle of comorbidities care — Pulmonary function tests, blood gas analysis, transthoracic echocardiography, sleep study after stabilization of patient's index clinical condition, thus 1 month after hospital discharge
  Arms: Intervention

SUMMARY:
The study will assess the potential benefit of implementing a complex bundle of interventions to treat important - often unrecognized - comorbidities in patients surviving an episode of Acute Hypercapnic Respiratory Failure (AHRF). This study will also provide a comparative analysis of the costs and health consequences of two alternative strategies to inform decision making about healthcare. All interventions are individually evidence-based and seem sound to hypothesize that implementing such interventions might improve patient's outcome and reduce the financial burder of repeated hospitalization in AHRF survivors.

ELIGIBILITY:
Inclusion Criteria:

* Consent form signed
* Acute hypercapnic respiratory failure defined as PaCO2 > 6.3 kPa requiring invasive or non-invasive mechanical ventilation in the ICU

Exclusion Criteria:

* Age < 18 years old
* Known or suspected neuromuscular diseases
* Pregnancy
* Iatrogenic respiratory failure (i.e. drug overdose, AHRF after starting opiates or increasing opiates dose)
* Life expectancy < 3 months
* Confusion or major psychiatric illness
* Patient unable to be weaned from NIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Hospital readmission | 1-year observation
  Hospital or ICU readmission

SECONDARY OUTCOMES:
Health Related Quality of Life | Measured at regular 3, 6 and 12 months visits following patient's hospital discharge
  Hospital Anxiety and Depression scale (0 to 21 points with 21 indicating higher levels of anxiety and depression) Saint George Questionnaire (0-100 with 100 indicating more limitations) Impact of dyspea on daily activities measured by mMRC (0 to IV with IV indication more impact of dyspnea)
Cost-effectiveness | 1-year observation
  Costs related to unplanned emergency visits and hospital length of stay following readmission

CONTACTS AND LOCATIONS:
Overall Officials: Dan Adler, MD, Principal Investigator — University Hospital, Geneva
Locations (3):
- Centre Hospitalier Universitaire Grenoble Alpes, Grenoble, France
- Switzerland (2):
  - Geneva University Hospitals, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne

IPD SHARING:
Plan to Share IPD: No